CLINICAL TRIAL: NCT03292848
Title: A Phase 1, Single-dose, Sequential Cohort, Nonrandomized Crossover Trial to Assess the Pharmacokinetics, Safety, and Tolerability of Oral Brexpiprazole in Children (6 to< 13 Years Old) With Central Nervous System Disorders
Brief Title: Trial to Assess the Pharmacokinetics, Safety, Tolerability of Oral Brexpiprazole in Children (6 to <13 Years Old) With Central Nervous System Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 331-201-00103
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: ADHD; Autism; Bipolar I Disorder; Conduct Disorder; Oppositional Defiant Disorder
Keywords: CNS Disorders; Brexpiprazole
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Conduct Disorder; Oppositional Defiant Disorder; Central Nervous System Diseases | interventions — brexpiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 to <13 Years of Age (Experimental): Two doses will be administered with a washout period of 14 days between the first dose of 1.5 mg the second dose of 3 mg.
  Interventions: Drug: Brexpiprazole
- 6 to <10 Years of Age (Experimental): Two doses will be administered with a washout period of 14 days between the first dose of 0.75 mg and the second dose of 1.5 mg.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Tablet
  Other Names: OPC-34712

SUMMARY:
A study to assess pharmacokinetics, safety and tolerability of brexpiprazole in children ages 6 to <13 years with CNS disorders.

DETAILED DESCRIPTION:
A US based nonrandomized, sequential cohort, crossover trial to assess pharmacokinetics, safety and tolerability of brexpiprazole in children ages 6 to <13 years with CNS disorders who are receiving antipsychotic treatment for their medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 6 and 12 years of age
* Subjects with CNS disorders including, but not limited to, ADHD, autism spectrum disorders, bipolar I disorder (subjects 10 to 12 years old only for bipolar), conduct disorder, oppositional defiant disorder, or any psychotic disorder and who are receiving antipsychotic treatment for their medical condition. Subjects' diagnoses will be determined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria and confirmed at screening using the Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL).
* Subjects must be considered psychiatrically/medically appropriate for participation in a clinical trial in which they will receive two doses of an antipsychotic medication.
* Subjects with good physical health, as determined by no clinically significant deviation from normal for all of the following, prior to enrollment in the trial:

  1. Medical history
  2. Clinical laboratory determination
  3. ECGs
  4. Physical examinations
* Subjects who are within the 5th to 95th percentile for gender-specific BMI for age from the Centers for Disease Control and Prevention growth charts and weight at least 15 kg (approx. 33 lbs)
* Ability to commit to remain fully abstinent or use 2 approved methods of birth control during the trial for 21 (± 2) days following the last dose of IMP for sexually active females of childbearing potential.
* Ability, in the opinion of the PI, of the subject and the subject's legally acceptable representative or caregiver(s) to understand the nature of the trial and follow protocol requirements, including all of the following:

  1. Comply with prescribed dosage regimens and tablet ingestion, as well as the discontinuation of prohibited concomitant medications
  2. Reliably return for scheduled visits
  3. To be reliably rated on assessment scales

Exclusion Criteria:

* Subjects with a clinical presentation or history that is consistent with delirium, dementia, amnesia, or other cognitive disorders; subjects with psychotic symptoms that are better accounted for by another general medical condition(s) other than those listed in the second inclusion criterion above, or direct effect of a substance (ie, medication, illicit drug use, etc.).
* Subjects with a history of at least mild intellectual disability as determined by IQ < 70, clinical evidence, or a social or school history that is suggestive of intellectual disability.
* Subjects who have any of the following:

  1. A significant risk of committing suicide based on history and the principal investigator's clinical judgment, or routine psychiatric status examination
  2. Current suicidal behavior
  3. Imminent risk of injury; active suicidal ideation
  4. Any lifetime history of suicidal behavior detected by the Children's Baseline/Screening version of the C-SSRS.
* Subjects with a lifetime history of a substance use disorder (as determined by the DSM-5 criteria), or current substance misuse including alcohol and benzodiazepines, but excluding caffeine and nicotine.
* Subjects who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV seropositive status/acquired immunodeficiency syndrome, or chronic hepatitis B or C. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not expose the subject to an undue risk of significant adverse event or interfere with assessments during the course of the trial.
* Subjects with insulin dependent diabetes mellitus (IDDM) are excluded. Subjects with non-IDDM may be eligible for the trial if their condition is determined to be stable.
* Subjects with epilepsy or a history of seizures (except for a single seizure episode, for instance childhood febrile seizure or post traumatic) or a history of severe head trauma or cerebrovascular disease (eg, stroke, transient ischemic attack, etc.).
* Any major surgery within 30 days prior to the first dose of IMP.
* Any history of significant bleeding or hemorrhagic tendencies.
* Blood transfusions within 30 days prior to first dose of IMP.
* Subjects with a positive drug screen for cocaine, marijuana (even if by prescription), or other illicit drugs, or alcohol are excluded and may not be retested or rescreened.
* Subjects who have supine or standing diastolic blood pressure, after resting for at least 5 minutes, ≥ 95 mmHg.
* Subjects who have had a dose of depot antipsychotics within 6 months of screening.
* Consumption of alcohol or grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to the first dose of IMP and throughout the trial
* Subjects who participated in a clinical trial and were exposed to IMP within the last 30 days prior to screening or who participated in more than 2 interventional clinical trials within the past year.
* Subjects with a history of neuroleptic malignant syndrome or hypersensitivity to atypical antipsychotics.
* Subjects with a history of true allergic (i.e. not intolerance) response to more than one class of medications.
* Subjects with a history of allergic reaction or a known or suspected sensitivity to any substance that is contained in the IMP formula.
* Subjects who do not tolerate venipuncture or have poor venous access that would cause difficulty for collecting blood samples.
* Prisoners or subjects who are compulsorily detained (e.g. juvenile detention, court-mandated treatment) for any reason.
* Inability to tolerate oral medication or swallow tablets.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) [PK] | Up to 22 days or early termination
  The maximum plasma concentration of drug will be assessed for brexpiprazole and its major metabolite DM-3411.
Area under concentration-time curve (AUC) calculated from time zero to time t (AUCt) [PK] | Up to 22 days or early termination
  AUCt will be assessed for plasma brexpiprazole and its major metabolite DM-3411 to determine average concentration of drug over time
AUC from time zero to infinity [PK] | Up to 22 days or early termination
  AUC infinity will be assessed for plasma brexpiprazole and its major metabolite DM-3411 to determine total drug exposure over time
Time of maximum plasma concentration (tmax) [PK] | Up to 22 days or early termination
  The amount of time that the maximum plasma concentration of drug will be assessed for plasma brexpiprazole and its major metabolite DM-3411
Terminal-phase elimination half-life (t½,z) [PK] | Up to 22 days or early termination
  t½,z will be assessed for plasma brexpiprazole and its major metabolite DM-3411 to determine drug persistence in the body
Apparent clearance of drug from plasma after extravascular administration (CL/F) [PK] | Up to 22 days or early termination
  CL/F for brexpiprazole only

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAES) [Safety] | Up to 22 days or early termination with a 21 day follow-up period
Clinical laboratory tests [Safety] | Up to 22 days or early termination
  Collect hematology, serum chemistry,and urinalysis will be assessed to determine the safety and tolerability of drug
Vital signs observed and change from baseline data (systolic and diastolic blood pressure) [Safety] | Up to 22 days or early termination
Vital signs observed and change from baseline data (heart rate) [Safety] | Up to 22 days or early termination
Vital signs observed and change from baseline data (respiratory rate) [Safety] | Up to 22 days or early termination
Vital signs observed and change from baseline data (body temperature) [Safety] | Up to 22 days or early termination
12-lead electrocardiogram (ECGs) [Safety] | Up to 22 days or early termination
Physical examinations (height) [Safety] | Up to 22 days or early termination
  Height is measured in cm,and will be used to calculate Body Mass Index (BMI)
Physical examinations (weight) [Safety] | Up to 22 days or early termination
  Weight is measured in kg, and will be used to calculate Body Mass Index (BMI)
Physical examinations- Body Mass Index (BMI) [Safety] | Up to 22 days or early termination
  Body Mass Index (BMI) measured using height (cm) and weight (kg)
Physical examinations- review of body systems [Safety] | Up to 22 days or early termination
  Subject will be examined by site staff for any notable changes
Simpson-Angus Scale (SAS) rating scale [Safety] | Up to 22 days or early termination
  Will be used in analysis of Extrapyramidal Symptoms (EPS)
Abnormal Involuntary Movement Scale (AIMS) [Safety] | Up to 22 days or early termination
  Will be used in analysis of Extrapyramidal Symptoms (EPS)
Barnes Akathisia Rating Scale (BARS) [Safety] | Up to 22 days or early termination
  Will be used in analysis of Extrapyramidal Symptoms (EPS)
Columbia-Suicide Severity Rating Scale (C-SSRS) [Safety] | Up to 22 days or early termination

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Alliance for Wellness dba Alliance for Research, Long Beach, California
  - New Hope Clinical Research, Charlotte, North Carolina
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Road Runner Research Ltd., San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah